CLINICAL TRIAL: NCT04298554
Title: Comparison of Cannabinoids to Placebo in Management of Arthralgia and Myofascial Pain Disorder of the Temporomandibular Region: A Randomized Clinical Trial.
Brief Title: Comparison of Cannabinoids to Placebo in Management of TMJ Pain and Myofascial Pain in the TMJ Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-07020513
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: TMJ Disorder; Myofacial Pain; TMD
Keywords: CBD; TMJ; TMD
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain | interventions — Cannabinoids; hempseed oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBD Oil (Experimental): CBD PURE CBD OIL 20mg/1ml concentration - 1 ml (20mg) qd PO, hold under tongue for 1 minute and swallow daily
  Interventions: Other: CBD Oil
- Placebo (hemp oil) (Placebo Comparator): CBD PURE Hemp Oil- 1 ml qd PO, hold under tongue for 1 minute and swallow daily
  Interventions: Other: Hemp Oil

INTERVENTIONS:
Other: CBD Oil — CBD PURE CBD OIL 20mg/1ml concentration
  Other Names: Cannabinoids
  Arms: CBD Oil
Other: Hemp Oil — CBD PURE HEMP OIL
  Arms: Placebo (hemp oil)

SUMMARY:
The aim of this study is to determine whether the cannabinoids taken orally in the form of cannabidiol (CBD oil-a major non-psychoactive component of marijuana) vs placebo (hemp oil) will provide pain relief and improved jaw function in those who suffer from either myofascial pain disorder and/or arthralgia of the temporomandibular region.

1. Primary Objectives To determine if the consumption of CBD oil is superior to placebo for the improvement in jaw pain.
2. Secondary Objectives To determine if the consumption of CBD oil is superior to placebo for the improvement in function of the temporomandibular joint.
3. Exploratory Objectives To determine if there are any adverse effects that result from the consumption of CBD oil or placebo.

DETAILED DESCRIPTION:
The United States National Institute of Health Survey in 2001 conducted a self-reported survey of 30,978 people and determined the overall prevalence of temporomandibular joint and muscles disorders to be 4.6%, with 6.3% women and 1.8% men [1]. Temporomandibular joint arthralgia which is often caused by inflammatory joint arthropathy [2] and is commonly seen in conjunction with myofascial pain of the masticatory region. Myofascial pain syndrome is classically characterized by focal areas of exquisite tenderness caused by trigger points. Temporomandibular joint arthralgia and myofascial pain disorder pertaining to the temporomandibular joint region will be defined according to the research diagnostic criteria below [3].

The exact mechanism of action of CBD is not fully understood and several mechanisms of action have been proposed. Studies have indicated that CBD acts on a system in humans called the endocannabinoid system comprised of the CB1 and CB2 receptors. CB receptors were found throughout the human body: CB1 receptors in the brain and CNS and CB2 receptors are found throughout the gut, spleen, liver, heart, kidneys, blood vessels, lymph cells, and reproductive organs. CB1 receptors in the CNS help maintain core functions such as motor activity, pain perception, stress response, and memory. CB2 receptors widely distributed throughout the body in peripheral organs serve as core components of the immune system, muscular system, and cardiovascular system [4]. The endocannabinoid system has physiological and pathophysiological roles in modulation of pain [5]. Petitet et al. (1998) found CBD considerably reduced the receptor activation of a potent classical CB1 receptor agonist. CBD has a very low affinity for both known cannabinoid receptors. However, CBD antagonizes CB1 and CB2 receptor agonists at doses considerably lower than those of CBD needed to activate cannabis receptors [6]. Pertwee et al. (2002) found CBD was also shown to display inverse agonism at the human CB2 receptor, which may be a rational basis for its anti-inflammatory properties [7]. Pertwee (2002) proposes that CBD also functions outside of CB1 and CB2 receptors. An endogenous cannabinoid, anandamide, produced anti-nociception through mechanisms outside of the endocannabinoid system acting on the vanilloid receptors. The vanilloid receptors may regulate the release of inflammatory molecules (substance P) following exposure to noxious stimuli playing a role in the transmission of pain signals [7]. This pathway is well studied in capsaicin (an active component of chili peppers). Capasicin can produce an analgesic effect by desensitizing the TRPV1 receptor (a vanilloid receptor) inhibiting substance P. CBD inhibits the uptake and hydrolysis of the endocannabinoid anandamide, thus increasing its concentration [8, 9]. CBD stimulates the vanilloid receptor type 1 (VR1) with a maximum effect similar in efficacy to that of capsaicin [8] without the side effect of burning sensation. Not all cannabinoid effects can be explained through the CB1 and CB2 receptors and their endogenous ligand, anandamide. Researchers investigated the mechanisms, by which CBD reduces inflammatory and neuropathic pain in animals [10]. They found that the cannabinoid-induced analgesic effect is absent in mice lacking glycine receptors and concluded that this receptor mediates suppression of chronic pain. In other mouse models, CBD binds to the GPR55 receptor, a putative cannabinoid receptor [11]. This effect is involved in the anti-inflammatory action of CBD. In human clinical trials, Blake (2005) assessed the efficacy and safety of cannabis-based medicine (Sativex) in the treatment of pain caused by rheumatoid arthritis. Sativex consists of a blend of plant extracts which delivers approximately equal amounts of THC and CBD. Statistically significant improvements in pain on movement, pain at rest, and quality of sleep [12]. The rationale for the starting dose is somewhat arbitrary, 600mg/2FL is the most popular with retail customers. It is the highest concentration available with the CBD PURE brand oil which allows study subjects to maximize on the possible benefits of CBD. Since there are little known side effects, the risk of a higher concentration of CBD causing more adverse side effects is minimal.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-70 years of age
* Ability to give informed consent
* Arthralgia of the temporomandibular joint as defined according to the RDC/TMD criteria (see below chart)[3] and/or Myofascial pain of masticatory muscles as defined according to the RDC/TMD criteria (see below chart)[3]
* Baseline pain must be greater than 3/10 as self-reported on the VAS

Exclusion Criteria:

* Allergy to study drug
* Traumatic injury of masticatory muscles or temporomandibular joint within last 12 months
* Mandibular fracture within last 12 months
* Pregnancy or breast feeding
* Initiation of additional treatment of MPD within the past 1 months
* Baseline pain less than 3/10 as self-reported on the VAS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2022-05-29 (Actual); Study Completion 2022-05-29 (Actual)

PRIMARY OUTCOMES:
Change in baseline in pain, as measured by the Visual Analog Scale (VAS) | Baseline, 3 weeks, 7 weeks, and 11 weeks
  Scores are measured from 1-100mm VAS. The VAS ranges from 0 to 100 with O indicating no pain and higher scores indicating a greater pain.

SECONDARY OUTCOMES:
Change in jaw functional limitations as measured by the jaw functional limitation scale. | Baseline, 3 weeks, 7 weeks, and 11 weeks
  Scores are measured from 5 (lowest) to 25 (highest). Higher scores reflect better jaw function.

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Reeve, DMD FACS, Principal Investigator — Weill Cornell New York Presbyterian Hospital
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No